CLINICAL TRIAL: NCT02764944
Title: Endoscopic Full Thickness Resection Without Exposure to Peritoneum: Single Center Single Arm Study
Brief Title: Endoscopic Full Thickness Resection Without Exposure to Peritoneum
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Chan Gyoo Kim, Senior Scientist, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2015-0171
Record Dates: First submitted 2016-04-08; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Submucosal Tumor of Stomach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): simple non-exposure EFTR group (single arm study)
  Interventions: Procedure: simple non-exposure EFTR

INTERVENTIONS:
Procedure: simple non-exposure EFTR — This intervention includes the steps of laparoscopic seromuscular suturing with a barbed suture thread (V-Loc), which results in inversion of the stomach wall; EFTR of the inverted stomach wall from inside the stomach; and finally, endoscopic mucosal suturing with endoloops and clips.

SUMMARY:
This study evaluates the feasibility of endo-laparoscopic full-thickness resection with simple suturing technique which did not expose gastric mucosa to peritoneum (simple non-exposure EFTR) in patients with gastric tumor.

DETAILED DESCRIPTION:
Current endoscopic full-thickness resection (EFTR) methods are limited by their transmural communication and exposure of tumor to peritoneum. Recently, endo-laparoscopic full-thickness resection with simple suturing technique which did not expose gastric mucosa to peritoneum (simple non-exposure EFTR) was developed. This new technique includes the steps of laparoscopic seromuscular suturing with a barbed suture thread (V-Loc), which results in inversion of the stomach wall; EFTR of the inverted stomach wall from inside the stomach; and finally, endoscopic mucosal suturing with endoloops and clips.

This study evaluates the feasibility of simple non-exposure EFTR technique in patients with gastric tumor. This study is single arm study and will be performed in single center.

ELIGIBILITY:
Inclusion Criteria:

* Gastric subepithelial tumor
* Tumor invades of muscularis propria on endoscopic ultrasonography (EUS) finding
* Tumor size more than 1.5cm or increasing size during observation

Exclusion Criteria:

* Tumor size more than 5cm
* Refuse to be enrolled to study.
* Bleeding tendency,
* Inappropriate condition for surgery with general anesthesia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
En bloc resection | During operation
  rate of en bloc resection (%)

SECONDARY OUTCOMES:
procedure time | During operation
  minutes
complication | 3 months
  leakage, re-operation, stenosis, etc.
successful closure of resection site | 1 week
  Rate of successful closure (%)

CONTACTS AND LOCATIONS:
Overall Officials: Chan G Kim, M.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No